CLINICAL TRIAL: NCT02387268
Title: Evaluation of the Performance of the "CleanC" System
Brief Title: Evaluation of the Performance of the CleanC System-Israel
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Motus GI Medical Technologies Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: CL00005
Record Dates: First submitted 2015-03-02; First posted 2015-03-12 (Estimated); Results first posted 2016-03-07 (Estimated); Last update posted 2017-09-20 (Actual); Status verified 2016-02

CONDITIONS: Colorectal Cancer (CRC) Screening
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CleanC (Experimental): Standard colonoscopy procedure using the CleanC system
  Interventions: Device: CleanC system

INTERVENTIONS:
Device: CleanC system — Cleansing liquid and fecal matter during a standard colonoscopy procedure

SUMMARY:
The Motus GI Colon Cleansing device is intended to facilitate intra-procedural cleaning of a poorly prepared colon by irrigating the colon and evacuating the irrigation fluid and feces.

DETAILED DESCRIPTION:
The study aim to evaluate the post Procedure Cleansing Level as Measured by the Boston Bowel Preparation Scale (BBPS).

Each subject was required to follow a bowel preparation regimen including split dose of 2 tablets of 5mg Bysacodyle followed by a colonoscopy procedure with the tested device.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects in the age range of 18-75 years
2. Subjects with BMI within the range of 18.5-35
3. Subject is willing to sign informed consent form

Exclusion Criteria:

1. Active or severe inflammatory bowel disease (IBD)
2. Subjects with severe diverticulitis \ diverticular disease (known or detected)
3. Known or detected colonic stenosis
4. Known or detected bowel obstruction
5. History of prior colon surgery
6. ASA≥IV (sever systemic disease)
7. Sever Renal insufficiency (Creatinine≥1.5mg%)
8. Sever Liver insufficiency (ALT/AST≥2UNL)
9. Contraindication for "colonoscopy" anesthesia \ sedation \ prep agent
10. pregnancy
11. Subjects with altered mental status/inability to provide informed consent
12. Subject has a condition or is in a situation which in the investigators opinion may put the subject at significant risk, may confound the study results, or may interfere significantly

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2015-05; Primary Completion 2015-06 (Actual); Study Completion 2015-11 (Actual)

IPD SHARING:
Plan to Share IPD: Undecided
De-identified individual participant for primary and secondary outcome measures may be become available in the future

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | CleanC
Started | 10
Completed | 9
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | CleanC
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.3 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 6
Region of Enrollment [Number; unit: participants]
  Israel | 10

OUTCOME MEASURES:

1. Primary Outcome: Percentage Subjects With Post Procedure Cleansing Level as Measured by the Boston Bowel Preparation Scale (BBPS) Adequate Cleansing-(BBPS>1 )
Description: Scale ranges- Min-0, Max-3 where:
  0 = Unprepared colon segment with mucosa not seen due to solid stool that cannot be cleared.
  1. = Portion of mucosa of the colon segment seen, but other areas of the colon segment not well seen due to staining, residual stool and/or opaque liquid.
  2. = Minor amount of residual staining, small fragments of stool and/or opaque liquid, but mucosa of colon segment seen well.
  3. = Entire mucosa of colon segment seen well with no residual staining, small fragments of stool or opaque liquid. The wording of the scale was finalized after incorporating feedback from three colleagues experienced in colonoscopy.
Time Frame: During the colonoscopy procedure withdrawal phase (10 min in average)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | CleanC
Number analyzed (Participants) | 9
percentage of participants | 88.9 [51.7 to 99.7]

2. Primary Outcome: Safety as Measured by Number of Serious Adverse Events and Major Complications.
Time Frame: Max of 9 days
Reporting Status: Not Posted

3. Secondary Outcome: Percentage of Participants in Whom the Cecum Was Reached
Description: A procedure was considered complete when the cecum was reached and visualized.
Time Frame: During the colonoscopy procedure
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | CleanC
Number analyzed (Participants) | 9
percentage of participants | 88.9 [51.7 to 99.7]

ADVERSE EVENTS:
Arm/Group | CleanC
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 1/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CleanC (N=10)
Mild abdominal pain (Gastrointestinal disorders) | 1 (1) — Mild abdominal pain was reports as probably related to colonoscopy procedure and not to Motus GI CleanC system

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No